CLINICAL TRIAL: NCT02695641
Title: A Phase 0 Study to Evaluate the Pharmacokinetics of Low-dose Bevacizumab and Its Efficacy on Reducing Plasma Free Vascular Endothelial Growth Factor-A (VEGF-A) in Hemodialysis Patients
Brief Title: Reduction of Plasma Free VEGF-A Using Low-dose Bevacizumab in Hemodialysis Patients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to enroll patients for the trial.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sanjay Misra, M.D., MD, Professor, Department of Radiology, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-007414
Record Dates: First submitted 2016-02-25; First posted 2016-03-01 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: End Stage Renal Disease; Hemodialysis Vascular Access Failure
Keywords: Arteriovenous Fistula; Arteriovenous Graft; Bevacizumab; Hemodialysis; VEGF; Avastin
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage 1 - Low dose administration (Experimental): Ten hemodialysis patients will receive IV infusion treatment with 1.25mg bevacizumab and undergo serial blood draws on Days 0, 1, 3, 6, 10, 15, 22, and 29 during dialysis sessions. ELISA will be performed to evaluate drug serum concentration and corresponding plasma free VEGF-A levels (pg/ml). The safety and pharmacokinetic/dynamic (PK/PD) data will be analysed and ≥50% VEGF-A suppression retained from baseline by Day 15 will be considered successful. If target outcomes are met in stage 1, the study will be terminated, otherwise the study will progress to stage 2.
  Interventions: Drug: 1.25mg bevacizumab
- Stage 2 - Dose escalation (Experimental): If outcomes are not met in stage 1, Ten additional hemodialysis patients will receive IV infusion treatment with 2.50mg bevacizumab treatment. They will undergo serial blood draws on Days 0, 1, 3, 6, 10, 15, 22, and 29 during dialysis sessions. ELISA will be performed to evaluate drug serum concentration and corresponding plasma free VEGF-A levels (pg/ml). The safety and PK/PD data will be analysed and ≥50% VEGF-A suppression retained from baseline by Day 15 will be considered successful. If target outcome is not met, the study will be terminated.
  Interventions: Drug: 2.50mg bevacizumab

INTERVENTIONS:
Drug: 1.25mg bevacizumab — Bevacizumab is a monoclonal antibody against VEGF-A. 1.25mg in 50ml 0.9% Sodium Chloride will be administered once as an intravenous infusion over 30 minutes.
  Other Names: Avastin
  Arms: Stage 1 - Low dose administration
Drug: 2.50mg bevacizumab — Bevacizumab is a monoclonal antibody against VEGF-A. 2.50mg in 50ml 0.9% Sodium Chloride will be administered once as an intravenous infusion over 30 minutes.
  Other Names: Avastin
  Arms: Stage 2 - Dose escalation

SUMMARY:
The primary purpose of this pilot study is to assess the pharmacokinetic profile of low-dose bevacizumab and its effectiveness in reducing plasma free VEGF-A levels safely in hemodialysis patients. This information will be used to plan a phase 1 clinical trial evaluating bevacizumab's role in hemodialysis vascular access failure.

DETAILED DESCRIPTION:
It has been found that hemodialysis arteriovenous fistula failure is partly mediated through a VEGF pathway. The administration of bevacizumab (a VEGF-A monoclonal antibody) in arteriovenous fistula (AVF) murine models at a dose of 5mg/kg (a standard chemotherapeutic dose) has shown a significant reduction in stenosis formation and an overall improvement in vascular remolding. However, previous pharmacokinetic human studies have shown that bevacizumab administered at a low dose of 1.25mg intravitreally (ocular neovascularization patients) is sufficient enough to suppress circulating VEGF-A levels up to 30 days post administration. A chart review on 14 hemodialysis patients receiving an arteriovenous access and intravitreal bevacizumab has demonstrated a significant improvement in patency (HR: 0.45, p-value: 0.037) when compared to controls. Prior to a phase 1 trial, it is essential to determine if intravenous administration of bevacizumab demonstrates the same pharmacokinetics and bio-response profile as intravitreal administration, and to determine the optimal dose and frequency. This phase 0 study will be conducted in 10 existing hemodialysis patients at a dose of 1.25mg with a potential dose escalation to 2.5mg if optimal results are not seen. The findings from this study can have a substantial clinical impact not only in ESRD patients but also in patients receiving other vascular or endovascular procedures.

ELIGIBILITY:
Inclusion Criteria

* Patients between 18 and 85 years old, inclusive
* Patients with end stage renal disease (ESRD) who are currently undergoing hemodialysis treatment through an upper extremity fistula
* Hemoglobin ≥8g/dL and platelet count ≥100,000/mm3 prior to Day 1
* Adequate liver function, defined as serum bilirubin ≤1.5 mg/dL; gamma-glutamyltransferase (GGT), aspartate aminotransferase (AST), alanine transaminase (ALT), and alkaline phosphatase ≤2x upper limit of normal or international normalized ratio (INR) ≤ 1.5 prior to Day 0 or INR ≤ 2 if on anticoagulant therapy.
* Ability to communicate meaningfully with investigative staff, competence to give written informed consent, and ability to comply with entire study procedures
* If female and of childbearing years, must have a negative serum pregnancy test at the screening visit (Visit 1). Both female patients of childbearing potential and male patients with childbearing potential partners must be willing to use contraception from the time of screening to completion of the study
* Life expectancy of at least 1 year

Exclusion Criteria

* Known sensitivity to bevacizumab or prior treatment with any medication known to target VEGF
* Current use of medications that are known to interact with the safety and efficacy of bevacizumab (most commonly: Antineoplastics (Anthracyclines), Belimumab, Bisphosphonate Derivatives, Clozapine, Dipyrone, Irinotecan, Sorafenib, and Sutent)
* History or evidence of severe cardiac disease (NYHA Functional Class III or IV), myocardial infarction within six months of study entry (Day 1), ventricular tachyarrhythmias requiring continuing treatment, or unstable angina
* Significant uncontrolled hypertension (systolic blood pressure above 160 mm Hg and/or diastolic blood pressure above 100 mm Hg);
* Stroke within six (6) months of study entry (Day 1)
* Treatment with any investigational drug/ device within 60 days prior to study entry (Day1)
* Treatment with vitamin K-antagonists or direct thrombin inhibitors with an INR ≥2
* All patients (including both female patients of childbearing potential and male patients with childbearing potential partners) who do not use a highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly), e.g. implants, injectables, combined oral contraceptives in combination with a barrier method, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner
* Malignancy or treatment for malignancy within the previous 6 months
* Immunodeficiency including AIDS / HIV or Active autoimmune disease
* Documented hypercoagulable state or history of 2 or more deep vein thromboses (DVTs) or other spontaneous intravascular thrombotic events
* Bleeding diathesis or Anemia with a hematocrit level of less than 30%
* A prothrombin time or a partial thromboplastin time more than 1.2 times the upper limit of normal, or absolute platelet counts below the lower limit of normal; an absolute neutrophil count below 1,500/mm3
* Active local or systemic infection (WBC > 15,000/mm3)
* Gastrointestinal ulcer or bleeding, or wound dehiscence
* Scheduled elective surgery within 2 months of start date
* Known serious allergy to aspirin or penicillin
* Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of bevacizumab
* Employees of the sponsor or patients who are employees or relatives of the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in Serum concentration of bevacizumab (nM) | baseline, 4 weeks
  Obtained through serial blood draws and measured through ELISA.
Change in plasma free VEGF-A levels (pg/ml) | baseline, 4 weeks
  Obtained through serial blood draws and measured through ELISA. ≥50% suppression from baseline retained by Day 15 will be considered successful.

SECONDARY OUTCOMES:
Safety Profile/ Adverse Events (NCI-CTCAE v. 4.0) monitoring | 4 weeks
  Monitoring of drug infusion reactions and adverse event development on subsequent follow-up visits at dialysis centers. Monitoring will include but will not be limited to allergic reactions or anaphylaxis, development of hypertension, excessive bleeding or thromboembolic events

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Misra, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang B, Janardhanan R, Vohra P, Greene EL, Bhattacharya S, Withers S, Roy B, Nieves Torres EC, Mandrekar J, Leof EB, Mukhopadhyay D, Misra S. Adventitial transduction of lentivirus-shRNA-VEGF-A in arteriovenous fistula reduces venous stenosis formation. Kidney Int. 2014 Feb;85(2):289-306. doi: 10.1038/ki.2013.290. Epub 2013 Aug 7. PMID 23924957
- [Background] Avery RL, Castellarin AA, Steinle NC, Dhoot DS, Pieramici DJ, See R, Couvillion S, Nasir MA, Rabena MD, Le K, Maia M, Visich JE. Systemic pharmacokinetics following intravitreal injections of ranibizumab, bevacizumab or aflibercept in patients with neovascular AMD. Br J Ophthalmol. 2014 Dec;98(12):1636-41. doi: 10.1136/bjophthalmol-2014-305252. Epub 2014 Jul 7. PMID 25001321
- [Background] Papadopoulos N, Martin J, Ruan Q, Rafique A, Rosconi MP, Shi E, Pyles EA, Yancopoulos GD, Stahl N, Wiegand SJ. Binding and neutralization of vascular endothelial growth factor (VEGF) and related ligands by VEGF Trap, ranibizumab and bevacizumab. Angiogenesis. 2012 Jun;15(2):171-85. doi: 10.1007/s10456-011-9249-6. PMID 22302382
- [Background] Matsuyama K, Ogata N, Matsuoka M, Wada M, Takahashi K, Nishimura T. Plasma levels of vascular endothelial growth factor and pigment epithelium-derived factor before and after intravitreal injection of bevacizumab. Br J Ophthalmol. 2010 Sep;94(9):1215-8. doi: 10.1136/bjo.2008.156810. Epub 2010 Jun 10. PMID 20538658
- [Background] Wang D, Choi KS, Lee SJ. Serum concentration of vascular endothelial growth factor after bilateral intravitreal injection of bevacizumab. Korean J Ophthalmol. 2014 Feb;28(1):32-8. doi: 10.3341/kjo.2014.28.1.32. Epub 2014 Jan 21. PMID 24505199
- [Background] Zehetner C, Kirchmair R, Huber S, Kralinger MT, Kieselbach GF. Plasma levels of vascular endothelial growth factor before and after intravitreal injection of bevacizumab, ranibizumab and pegaptanib in patients with age-related macular degeneration, and in patients with diabetic macular oedema. Br J Ophthalmol. 2013 Apr;97(4):454-9. doi: 10.1136/bjophthalmol-2012-302451. Epub 2013 Feb 5. PMID 23385630
- [Background] Garnier-Viougeat N, Rixe O, Paintaud G, Ternant D, Degenne D, Mouawad R, Deray G, Izzedine H. Pharmacokinetics of bevacizumab in haemodialysis. Nephrol Dial Transplant. 2007 Mar;22(3):975. doi: 10.1093/ndt/gfl664. Epub 2006 Nov 8. No abstract available. PMID 17093010
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials